CLINICAL TRIAL: NCT00529750
Title: Comparative Trial of the Effects of Irbesartan vs Atenolol on the Endothelial Function of Hypertensive Patients With Metabolic Syndrome
Brief Title: Effect of the Angiotensin II Receptor Antagonist Irbesartan on Biochemical and Functional Markers of Endothelial Dysfunction in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_8261
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Irbesartan; Atenolol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Irbesartan Group (Experimental): 150 mg p.o. once a day, 30 minutes before breakfast during 12 weeks
  Interventions: Drug: IRBESARTAN
- Atenolol Group (Active Comparator): 50 mg p.o. once a day, 30 minutes before breakfast during 12 weeks.
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: IRBESARTAN — Tablets
  Arms: Irbesartan Group
Drug: Atenolol — Tablets
  Arms: Atenolol Group

SUMMARY:
Primary:

* To evaluate the impact of irbesartan on endothelial function in hypertensive patients with metabolic syndrome.

Secondary:

* To evaluate the oxidative stress status in patients with hypertension with metabolic syndrome.
* To correlate the oxidative stress status with endothelial function in these patients.
* To evaluate the effect of irbesartan on the oxidative stress stage in patients with metabolic syndrome and to correlate it with the effect on endothelial function .
* To correlate the change in endothelial function and oxidative stress stage with the change of arterial pressure levels.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension grade 1 or 2
* With at least two of the following criteria for the diagnosis of metabolic syndrome:

  * Body mass index > or = 25 kg/m2 AND waist circumference > or = 100 cm.
  * Dyslipidemia (triglycerides fasting serum levels > or = 200 mg/dL OR HDL serum levels < or = 40 mg/dL)
  * Fasting serum glucose > or = 110 mg/dL but < 126 mg/dL

Exclusion Criteria:

* Known hypersensitivity to Irbesartan
* Hypertension grade 3
* History of clinical vascular events such as TIAs, stroke, peripheral arterial disease
* Coronary artery disease
* Renal insufficiency (creatinine serum levels > or = 1.2 mg/dL)
* Presence of clinical heart failure
* Asthma and COPD
* Valvular cardiopathy clinically relevant
* Current therapy with antioxidant drugs, statins
* Therapy with AIIRA for at least 3 months during the last semester
* Presence of any acute illness or major trauma in the last 8 weeks
* History of a chronic inflammatory disease such as rheumatoid arthritis, immune disorders or connective tissue disease.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2002-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function in vivo qualification: brachial artery flow mediated vasodilation (FMV%) determined by high resolution ultrasound. | at baseline and at the end of the study-12th wk

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Gomez, Study Director — Sanofi